CLINICAL TRIAL: NCT06429514
Title: Based on the Theory of Gut-brain Axis, the Intervention Effect and Related Mechanism of Ganoderma Lucidum Spore Powder on Depressive Symptoms in Patients With Thyroid Cancer Were Investigated
Brief Title: Study on the Mechanism of Ganoderma Lucidum Spore Powder in the Treatment of Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ling Zhiqiang (Other)
Collaborators: Zhejiang Shouxiangu Pharmaceutical Co,. Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Ling Zhiqiang, Principal Investigator, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2023-307
Record Dates: First submitted 2024-05-15; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Depression; Thyroid Cancer
Keywords: Depression; Thyroid Cancer; the gut-brain axis; ganoderma lucidum
MeSH Terms: conditions — Depression; Thyroid Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients with depressive symptoms after papillary thyroid carcinoma surgery 300 cases ; there were 200 cases in the experimental group and 100 cases in the control group. From the first day after enrollment, the subjects were given 4 g of the test drug ( Ganoderma lucidum spore powder or placebo ) every day for 90 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ganoderma lucidum spore powder (Experimental): Oral administration of Ganoderma lucidum spore powder 4g per day ( 1 bag at a time, 2 times a day, 2g / bag ) for 90 days
  Interventions: Dietary Supplement: Ganoderma lucidum spore powder
- placebo (Placebo Comparator): Oral ' placebo ' 4g per day ( 1 bag at a time, 2 times a day, 2g / bag ) for 90 days.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: Ganoderma lucidum spore powder — One bag at a time, 2 times a day, 2g / bag
  Arms: Ganoderma lucidum spore powder
Other: placebo — One bag at a time, 2 times a day, 2g / bag
  Arms: placebo

SUMMARY:
To clarify the clinical effect of Ganoderma lucidum spore powder intervention on postoperative depressive symptoms of papillary thyroid carcinoma ; to elucidate the antidepressant mechanism of Ganoderma lucidum spore powder.

DETAILED DESCRIPTION:
After being informed of the study and potential risks, all patients who gave written informed consent were enrolled. A total of 300 eligible patients were randomly assigned in a double-blind manner and divided into experimental group and control group at a ratio of 2 : 1. The subjects were given oral test drugs ( Ganoderma lucidum spore powder or placebo ) 4g per day for 90 days from the first day after enrollment.

ELIGIBILITY:
Inclusion Criteria

* patients with depressive symptoms after surgery for papillary thyroid carcinoma in the outpatient department of Zhejiang Cancer Hospital
* Han nationality
* No previous depression and other mental diseases
* 18-80 years old
* Women
* BMI 19 ~ 24

Exclusion Criteria

* suffering from other diseases of the intestinal system
* Gastrointestinal surgery was performed before intervention
* Including patients with other malignant tumors, who need chemotherapy, radiotherapy, biological therapy or traditional Chinese medicine treatment received antibiotics or microecological modulators within 3 months before the intervention
* Acute intestinal obstruction
* Patients with severe depressive symptoms who must receive antidepressant treatment organic diseases such as heart and brain diseases, brain trauma history of mental illness, use of psychoactive drugs such as drugs
* Severe liver and kidney dysfunction
* Pregnancy, lactation

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-05-03 (Actual)

PRIMARY OUTCOMES:
Depression symptoms relieved | Day0,Month3
  hamilton depression rating scale relieved from 8-20 to ≤8

SECONDARY OUTCOMES:
Changes of intestinal microbial diversity in patients | Day0,Month3
  The increase of intestinal microbial diversity and abundance

CONTACTS AND LOCATIONS:
Overall Officials: Jinbiao Shang, Study Director — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/14/NCT06429514/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/14/NCT06429514/ICF_001.pdf